CLINICAL TRIAL: NCT06316427
Title: Autologous and Donor-derived CD7 CAR T-cell Therapy in Refractory or Relapsed T-cell Malignancies: a Multi-center, Open-label, Phase Ⅰ/Ⅱ Clinical Trial
Brief Title: Autologous and Donor-derived CD7 CAR-T Therapy in Refractory or Relapsed T-cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: The General Hospital of Western Theater Command (Other); Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai (Other); Shanghai Liquan Hospital (Other); Central People's Hospital of Zhanjiang (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2024-003
Record Dates: First submitted 2024-03-08; First posted 2024-03-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-03

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia, in Relapse; Refractory Acute Lymphoblastic Leukemia; T-cell Malignancies
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Investigator Initiate Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm-1 (Experimental): Autologous CD7 CAR T-cell treatment
  Interventions: Drug: Autologous CD7 CAR T-cell
- Arm-2 (Experimental): Prior-HSCT donor-derived CD7 CAR T-cell treatment
  Interventions: Drug: Prior-HSCT donor-derived CD7 CAR T-cell
- Arm-3 (Experimental): New donor-derived CD7 CAR T-cell treatment
  Interventions: Drug: New donor-derived CD7 CAR T-cell

INTERVENTIONS:
Drug: Autologous CD7 CAR T-cell — Peripheral blood mononuclear cells for the production of CD7 CAR T cells are collected from patients.
  Arms: Arm-1
Drug: Prior-HSCT donor-derived CD7 CAR T-cell — Peripheral blood mononuclear cells for the production of CD7 CAR T cells are collected from prior-HSCT donors.
  Arms: Arm-2
Drug: New donor-derived CD7 CAR T-cell — Peripheral blood mononuclear cells for the production of CD7 CAR T cells are collected from new donors.
  Arms: Arm-3

SUMMARY:
This is a multi-center, open-label, non-randomized, phase I/II trial. Patients with refractory or relapsed T-cell malignancies will receive autologous, prior-HSCT donor-derived or new donor-derived CD7 CAR T cells according to their HSCT history, peripheral blood leukemia burden and at their discretion. The primary objective is to learn about the safety of autologous, prior-HSCT donor-derived and new donor-derived CD7 CAR T-cell therapy in patients with refractory or relapsed T-cell acute lymphoblastic leukemia and lymphoma (r/r T-ALL/T-LBL) in phase I and to learn about the efficacy of autologous, prior-HSCT donor-derived and new donor-derived CD7 CAR T-cell therapy in patients with refractory or relapsed T-cell acute lymphoblastic leukemia and lymphoma (r/r T-ALL/T-LBL) in phase II. The primary endpoint is type and incidence of dose limiting toxicity (DLT) within 21 days after CD7 CAR T-cell infusion in phase I and overall response rate (ORR), which includes CR, CRh, CRi, MLFS, aplastic marrow for blood and bone marrow; central nervous system (CNS) remission; CR and PR for lymphomatous extramedullary disease according to National Comprehensive Cancer Network (NCCN) Guidelines Version 3.2023 of Acute Lymphoblastic Leukemia at 3 months (± 1 week) post CD7 CAR T-cell infusion in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells in phase II. A total number of 80 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Only patients who meet all the following criteria can be included in the group:

1. CD7-positive refractory or relapsed T-cell malignancies with progression or intolerance after all standard treatments, limited prognosis from currently available treatments and no available treatment options (e.g. HSCT or chemotherapy).
2. Tumor cells in bone marrow or cerebrospinal fluid are positive for CD7 antigen by flow cytometry or tumour tissue is positive for CD7 by immunohistochemistry (CD7 antigen positivity by flow cytometry: >80% of tumour cells expressing CD7 with a mean fluorescence intensity [MFI] of CD7 similar to that of normal T cells are considered to have fully positive expression; >80% of tumor cells expressing CD7 but with an MFI of CD7 at least 1 log lower than that of normal T cells are considered to have low expression [dim]; tumor cells with a CD7 expression rate between 20-80% are considered to have partial expression; CD7 antigen positivity by pathological immunohistochemistry: >30%);
3. Male or female, age 1-70 years;
4. No severe allergic constitution;
5. Eastern Cooperative Oncology Group (ECOG) performance status score (Oken et al., 1982) of 0-2;
6. Life expectancy of at least 60 days as determined by the investigator;
7. Provide a signed informed consent form prior to any screening procedures; subjects volunteering to participate in the study should be capable of understanding and signing the informed consent form and be willing to follow the study visit schedule and associated study procedures as specified in the protocol. Subjects aged 19-70 years old need to be sufficiently aware and capable of signing the informed consent form; subjects aged 1-7 years can be recruited after legal guardians or patient advocates sign the informed consent form; subjects aged 8-18 years need to be sufficiently aware and able to sign the informed consent form, and their legal guardians or patient advocates also need to sign the informed consent form.

Exclusion Criteria:

Patients with at least one of the following conditions are excluded:

1. Intracranial hypertension or unconscious;
2. Acute heart failure or severe arrhythmia;
3. Acute respiratory failure;
4. Other types of malignant tumors;
5. Diffuse intravascular coagulation;
6. Serum creatinine and/or blood urea nitrogen over 1.5 times the normal value;
7. Sepsis or other uncontrolled infection;
8. Uncontrolled diabetes mellitus;
9. Severe psychological disorder;
10. Obvious cranial lesions by cranial MRI;
11. Allergic constitution;
12. Organ recipients;
13. Pregnant or breastfeeding;
14. Active, uncontrolled infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or treponema pallidum (TP).

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) in phase I | 21 days post infusion
  Type and incidence of dose-limiting toxicity (DLT) within 21 days after CD7 CAR T-cell infusion
Overall Response Rate (ORR) in phase II | 3 months (± 1 week) post infusion
  Overall response rate (ORR), which includes CR, CRh, CRi, MLFS, aplastic marrow for blood and bone marrow; central nervous system (CNS) remission; CR and PR for lymphomatous extramedullary disease per National Comprehensive Cancer Network (NCCN) Guidelines Version 3.2023 of Acute Lymphoblastic Leukemia at 3 months (± 1 week) post CD7 CAR T-cell infusion in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells

SECONDARY OUTCOMES:
Overall Response Rate (ORR) in phase I | 3 months (± 1 week) post infusion
  Overall response rate (ORR), which includes CR, CRh, CRi, MLFS, aplastic marrow for blood and bone marrow; central nervous system (CNS) remission; CR and PR for lymphomatous extramedullary disease per National Comprehensive Cancer Network (NCCN) Guidelines Version 3.2023 of Acute Lymphoblastic Leukemia at 3 months (± 1 week) post CD7 CAR T-cell infusion in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells
Safety in phase II | 2 years post infusion
  The adverse events in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells will be assessed according to the 2019 Consensus on Cytokine Release Syndrome and Immune-cell-associated Neurotoxicity published by the American Society of Transplantation and Cell Therapy (ASTCT), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and EBMT 2019 consensus.
Progression-Free Survival (PFS) in phase II | 2 years post infusion
  Progression-free survival (PFS) in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells.
Duration of Remission (DOR) in phase II | 2 years post infusion
  Duration of remission (DOR) in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells.
Overall Survival (OS) in phase II | 2 years post infusion
  Overall survival (OS) in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells.
Levels of CD7 CAR-T Cells in phase II | 2 years post infusion
  Levels of CD7 CAR-T cells in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells
Levels of CAR transgene in phase II | 2 years post infusion
  Levels of CAR transgene in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells
Levels of immune cells in phase II | 2 years post infusion
  Levels of immune cells in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells
Levels of cytokines in phase II | 2 years post infusion
  Levels of cytokines in refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma (r/r T-ALL/T-LBL) patients treated with CD7 CAR T cells

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - Shanghai Liquan Hospital, Shanghai, Shanghai Municipality
  - The General Hospital of Western Theater Command PLA, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No